CLINICAL TRIAL: NCT05041686
Title: A Prospective, Multi-site, Single Cohort, Non-controlled, Non-randomized Clinical Trial Evaluating the Usefulness of CADISS® System for the Cleavage of Severe Adhesions in Acute Cholecystitis (Cholecystectomy)
Brief Title: Usefulness of the CADISS® System for the Cleavage of Severe Adhesions in Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AuXin Surgery SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CADISS1703
Record Dates: First submitted 2021-09-01; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-08

CONDITIONS: Cholecystitis, Acute
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CADISS® System (Experimental)
  Interventions: Combination Product: CADISS® System

INTERVENTIONS:
Combination Product: CADISS® System — The CADISS® device was procured from AuXin Surgery. It consists in three elements:
  1. A single use disposable Remote Kit, containing a sterile cartridge, which prepares the Drug Product immediately before use, and the sterile tubing for fluid connexion. The Drug Product is a 30 ml sterile 5% mesna solution of pH 7.3+/-0.5 2.
  2. Reusable stainless steel noncutting mechanical instruments similar to those used in the normal practice, except for the provision of an internal irrigation channel bringing the Drug Product at the working edge.
  3. A pedal controlled electric motor driving the peristaltic cassette included in the disposable tubing in order to control the dispensing of the Drug Product during the procedure.

SUMMARY:
Acute cholecystitis is the most common complication of cholelithiasis. Acute cholecystitis is inflammation of the gallbladder that develops over hours, usually due to an obstruction of the cystic duct by a gallstone. Removal of the gallbladder (Cholecystectomy) is the only definitive treatment for acute cholecystitis, with laparoscopic cholecystectomy (LC) considered the gold standard. Serious complications that may occur with laparoscopic cholecystectomy, including bile duct injury, bile leaks, bleeding, and bowel injury, result in part from the anatomy, disease related pathology and structural misidentification due to inflammatory process (Gupta 2019).

The CADISS® System, Chemically Assisted mechanical DISSection, is intended for the selective detachment of pathological tissue layers and/or fibrotic tissues in various surgical procedures without using cutting instruments. It is based on the property of the drug mesna (Sodium 2-mercaptoethane sulfonate) to cleave the disulfide bonds responsible for the adherence of pathological tissues and for the strength of fibrosis. This study is a prospective, multi-sites, open label, single cohort clinical trial evaluating the use of CADISS® system to facilitate dissection of severe adhesions in cholecystectomy and to allow better identification of different structure.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Weight > 30 kg
* Confirmed diagnosis of acute gallstone cholecystitis
* Symptomatic or asymptomatic cholecystitis
* Under surgery for cholecystectomy:
* for the 5 first patients : cholecystectomy will take place within 72 hours of the first symptoms of cholecystitis
* after the 5 first patients : cholecystectomy will be allowed at any time after the first symptoms and at physician judgment
* Patient agrees to signed the informed consent

Exclusion Criteria:

* < 18 years old
* ≤ 30 kg
* Known hypersensibility to mesna
* Patient taking anticoagulant at the screening visit
* Patient having a pancreatitis or angiocholitis
* Patients suffering from hepatic or renal disorders
* Unable to sign the informed consent
* Participation in any study involving an investigational drug or device within the past 3 Months.
* Patient is pregnant, breastfeeding or has wish of pregnancy during the study.
* Individuals under tutorship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Ability of the CADISS® System to dissect adherences without cutting | Surgery
  Percentage of successful dissection

SECONDARY OUTCOMES:
The facilitation of detachment with the CADISS System | Surgery
  Likert scale - 0 to 10, the parameter is evaluated in comparison to the current surgeon practice. A score of 5 representing an appreciation of equivalence for the parameter with the current practice
The change of bleeding with the use of the CADISS System | Surgery
  Likert scale - 0 to 10, the parameter is evaluated in comparison to the current surgeon practice. A score of 5 representing an appreciation of equivalence for the parameter with the current practice. A score above 5 means the use of CADISS System reduction reduce bleeding compared to the current practice.
A change of surgical complication risk | Surgery
  Likert scale - 0 to 10, the parameter is evaluated in comparison to the current surgeon practice. A score of 5 representing an appreciation of equivalence for the parameter with the current practice. A score above 5 means the use of the CADISS System reduce the risk of surgical complication risks compared to the current practice.
The capability of the CADISS System to highlight the cleavage plane | Surgery
  Likert scale - 0 to 10, the parameter is evaluated in comparison to the current surgeon practice. A score of 5 representing an appreciation of equivalence for the parameter with the current practice. A score above 5 means an improvement compared to the current practice
The ease of use of the CADISS System | Surgery
  Likert scale - 0 to 10, A score of 0 representing the worse outcome
The easiness of control of the topical application with the CADISS System | Surgery
  Likert scale - 0 to 10, A score of 0 representing the worse outcome
Adverse events | Surgery, 2 to 5 days after surgery (Hospital discharge), 6 weeks follow-up
  All CADISS® related adverse events will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse Lubansu, Principal Investigator — University Hospital Erasme, Brussels, Belgium
Locations (1):
- AuXin Surgery, Louvain-la-Neuve, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malvaux P, Gherardi D, Gryspeerdt F, De Gheldere C. The utility of the CADISS(R) system in laparoscopic cholecystectomy for acute cholecystitis. Surg Endosc. 2022 Dec;36(12):9462-9468. doi: 10.1007/s00464-022-09616-w. Epub 2022 Nov 1. PMID 36319896